CLINICAL TRIAL: NCT02526277
Title: A Randomized Prospective Study on the Efficacy of the MMF07 Foot Massager and Heat Therapy Treatments for Restless Leg Syndrome
Brief Title: A Study on the Use of the MMF07 Foot Massager and Heat Therapy Treatments for Restless Leg Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariane Park (Other)
Collaborators: MedMassager (Unknown)
Responsible Party: Sponsor-Investigator, Ariane Park, MD, MPH, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2015H0107
Record Dates: First submitted 2015-07-22; First posted 2015-08-18 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Restless Legs Syndrome
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Diathermy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- MMF07 Foot Massager device (Active Comparator): Participants randomized to the MMF07 Foot Massager device arm will be provided the MMF07 Foot Massager device and instructed to set this device at setting 3, then increase or decrease the setting to their desired level of comfort, to be used for 30 minutes at bedtime.
  Interventions: Device: MMF07 Foot Massager
- Heat therapy (Active Comparator): Participants randomized to heat therapy will be provided an electric heating pad and will be instructed to use this pad at a medium setting for 30 minutes at bedtime.
  Interventions: Device: Heat Therapy
- MMF07 Foot Massager device and heat therapy (Active Comparator): Participants randomized to both the MMF07 Foot Massager device and heat therapy will be provided both the MMF07 Foot Massager device and electric heating pad. Participants will be instructed to set the MMF07 Foot Massager device at setting 3, then increase or decrease the setting to their desired level of comfort. They will also be instructed to use the electric heating pad at a medium setting at the same time for 30 minutes at bedtime.
  Interventions: Device: MMF07 Foot Massager; Device: Heat Therapy
- No treatment (No Intervention): Participants receiving no intervention will be asked to not alter their nighttime routine.

INTERVENTIONS:
Device: MMF07 Foot Massager
  Arms: MMF07 Foot Massager device; MMF07 Foot Massager device and heat therapy
Device: Heat Therapy
  Arms: Heat therapy; MMF07 Foot Massager device and heat therapy

SUMMARY:
The purpose of this study is to assess whether the MMF07 Foot Massager and/ or heat therapy may improve symptoms of restless legs syndrome (RLS). It will also assess the effect of the MMF07 Foot Massager and/ or heat on quality of life and sleep in people affected by RLS. Participants will be randomly assigned to one of four treatment groups;

1. MMF07 Foot Massager device
2. Heat therapy
3. Heat therapy and the MMF07 Foot Massage device
4. Neither heat nor MMF07 Foot Massager device (no treatment group)

DETAILED DESCRIPTION:
Few clinical trials have looked into non-pharmacological, non-invasive treatments for restless legs syndrome, despite reports that massage, baths and vibrations can alleviate RLS symptoms. We would like to assess whether the MMF007 Foot Massager device and/or heat therapy is associated with improved severity of RLS symptoms.

For this study the investigator will enroll 40 participants who have been diagnosed with restless legs syndrome, who will be followed over the course of four weeks and asked to complete two in person study visits. In the study the investigator is comparing the use of the MMF007 Foot Massager device and/ or heat therapy to a non treatment group to assess if the symptoms of RLS improve.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18-75 years old diagnosed with RLS according to the diagnostic criteria of the International Restless Legs Syndrome Study Group (11)
2. Subjects should have bothersome RLS symptoms, despite best medical therapy
3. Subjects should be stable on all RLS medication for at least 4 weeks prior to enrollment
4. All subjects must have vision and be proficient in English for compliance with testing and surveys
5. All women of childbearing age must be using an acceptable form of birth control, including abstinence, intrauterine device (IUD) or intrauterine system in place for at least 3 months prior to screening, subject or partner using barrier method (e.g., condom, diaphragm, or cervical cap) with spermicide from screening through study completion; partner has a documented vasectomy > 6 months prior to Baseline, Stable hormonal contraception (with approved oral, transdermal, or depot regimen) for at least 3 months prior to screening

Exclusion Criteria:

1. RLS secondary associated with end stage renal disease, iron deficiency or pregnancy
2. Concomitant sleep disorders
3. Any other condition (other than the primary indications), which in the opinion of the investigators might contribute to difficulty complying with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Park, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MMF07 Foot Massager Device: Participants randomized to the MMF07 Foot Massager device arm will be provided the MMF07 Foot Massager device and instructed to set this device at setting 3, then increase or decrease the setting to their desired level of comfort, to be used for 30 minutes at bedtime.
  MMF07 Foot Massager
- Heat Therapy: Participants randomized to heat therapy will be provided an electric heating pad and will be instructed to use this pad at a medium setting for 30 minutes at bedtime.
  Heat Therapy
- MMF07 Foot Massager Device and Heat Therapy: Participants randomized to both the MMF07 Foot Massager device and heat therapy will be provided both the MMF07 Foot Massager device and electric heating pad. Participants will be instructed to set the MMF07 Foot Massager device at setting 3, then increase or decrease the setting to their desired level of comfort. They will also be instructed to use the electric heating pad at a medium setting at the same time for 30 minutes at bedtime.
  MMF07 Foot Massager
  Heat Therapy
Period: Overall Study
Arm/Group | MMF07 Foot Massager Device | Heat Therapy | MMF07 Foot Massager Device and Heat Therapy | No Treatment
Started | 8 | 6 | 7 | 7
Completed | 8 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMF07 Foot Massager Device | Heat Therapy | MMF07 Foot Massager Device and Heat Therapy | No Treatment | Total
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 28
Age, Continuous [Median (Full Range); unit: years] | 65.8 [36.5 to 73.1] | 59.6 [55.6 to 72.8] | 59.9 [34.9 to 72.4] | 52.7 [39.2 to 70.2] | 59.6 [34.9 to 73.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 5 | 4 | 19
  Male | 1 | 3 | 2 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 6 | 7 | 7 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Married [Count of Participants; unit: Participants] — Number of participants who classified themselves as being married while enrolled in the study.
  Participants | 3 | 0 | 2 | 3 | 8
RLS Severity [Count of Participants; unit: Participants] — The severity of restless legs syndrome discomfort is measured by using the International Restless Legs Severity Scale. It is a 40 point scale measuring severity of restless leg symptoms. Patients are asked to answer a series of 10 questions each of which have values ranging from 0 to 4 and the points are then added. Higher values are associated with more severe symptoms.
  Participants
    Mild/moderate | 4 | 3 | 4 | 3 | 14
    Severe/very severe | 4 | 3 | 3 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: The International Restless Legs Severity Scale
Description: Participants answer a series of 10 questions each of which have values ranging from 0 to 4, the points are then added together. Higher values are associated with more severe symptoms; up to a maximum severity score of 40 points and a minimum severity of 0 points.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- No Treatment: Participants who received no intervention
Arm/Group | Heat Therapy | MMF07 Foot Massager Device | MMF07 Foot Massager Device and Heat Therapy | No Treatment
Number analyzed (Participants) | 6 | 8 | 7 | 7
score on a scale | 17.3 (8.1) | 12.3 (4.2) | 16.9 (6.2) | 21.3 (8.5)

2. Secondary Outcome: The Restless Legs Quality of Life Questionnaire
Description: Participants answer a series of 18 questions that are scored such that lower scores indicate worse quality of life. The scoring process for the RLSQoL is relatively complicated. Items 1-5, 7-10, and 13 use scales ranging from 1 to 5, with lower scores indicating a greater frequency and interference of restless legs syndrome. The total score for these items is converted to a value between 0 and 100 using an algorithm provided along with the scale. Items 6 and 16-18 require respondents to indicate how many days in the previous month or hours in the previous day they have been able to complete certain activities or have had their daily functioning interfered with. These items are scored as continuous variables (for example, ranging from 0 to 28 days for questions regarding the number of days per month). Items 11, 12, 14, and 15 are categorical variables, where a response of "yes" receives (a 1), a response of "no" receives (a 2), and a response of "not applicable receives (3a).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- No Treatment: Participants received no intervention
Arm/Group | MMF07 Foot Massager Device | Heat Therapy | MMF07 Foot Massager Device and Heat Therapy | No Treatment
Number analyzed (Participants) | 8 | 6 | 7 | 7
score on a scale | 82.4 (20.9) | 66.7 (25.6) | 74.2 (19.1) | 57.1 (32.6)

3. Secondary Outcome: Changes in Sleep as Measured by the Medical Outcomes Sleep Study Scale at Week 4
Description: Participants answered a series of 12 questions assessing sleep, with values ranging from 1 to 6, and an additional dichotomous indicator of optimal sleep. All items are scored so that a high score reflects more of the attribute implied by the scale name. Each item is then converted to a 0 to 100 possible range so that the lowest and highest possible scores are set at 0 and 100, respectively. In this format, scores represent the achieved percentage of the total possible score. Reference: Spritzer, K. L. & Hays, R. D. (2003, November). MOS Sleep Scale: A Manual for Use and Scoring, Version 1.0. Los Angeles, CA.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMF07 Foot Massager Device | Heat Therapy | MMF07 Foot Massager Device and Heat Therapy | No Treatment
Number analyzed (Participants) | 8 | 6 | 7 | 7
score on a scale | 26.6 (9.9) | 31.2 (15.8) | 37.0 (3.7) | 48.6 (18.4)

ADVERSE EVENTS:
Time Frame: Participants were seen at a Baseline visit and then followed up approximately 4 weeks later for a maximum of 31 days participation.
Arm/Group | MMF07 Foot Massager Device | Heat Therapy | MMF07 Foot Massager Device and Heat Therapy | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 0/6 | 4/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMF07 Foot Massager Device (N=8) | Heat Therapy (N=6) | MMF07 Foot Massager Device and Heat Therapy (N=7) | No Treatment (N=7)
Tingling (Nervous system disorders) | 0 (0) | 0 | 1 (1) | 0 — Tingling in bilateral feet
influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — migraine headache
itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — intermittent itching of bilateral feet and ankles
sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
jerking (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — right leg jerking
itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — bilateral itching on bottom of each foot
neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — worsening of neuropathy
low folic acid level (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02526277/Prot_SAP_000.pdf